CLINICAL TRIAL: NCT01001039
Title: Validation of the FAcial and CEphalic PAin INventory (FACE PAIN)
Brief Title: Validation of the Facial and Cephalic Pain Inventory
Acronym: FACE PAIN
Status: Completed | Type: Observational
Sponsor: Greg Davis (Other)
Responsible Party: Sponsor-Investigator, Greg Davis, Assistant Professor, University of Washington
Organization: University of Washington (Other)
Other Study IDs: 37055-E/A
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Sinusitis
Keywords: chronic sinusitis; facial pain
MeSH Terms: conditions — Sinusitis; Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: Patients seen in the Otology clinic who have not had sinus surgery in the past 2 months or a history of sinusitis in the last 6 months.
- cases: Patients seen in the Rhinology Clinic with a complaint of facial pain. They must have evidence of chronic sinusitis.

SUMMARY:
This study proposes to develop and validate a new instrument designed to measure facial and nasal discomfort related to chronic sinusitis. The second phase of the study will be to use this instrument to measure correlation with sinus computed tomography (CT) scans.

DETAILED DESCRIPTION:
The following specific aims will be addressed:

* to create a user-friendly, self-explanatory instrument (FACE PAIN questionnaire) with pain severity visual analog scales associated with the common locations of facial pain in chronic sinusitis.
* to evaluate the clinimetric reliability and validity of the FACE PAIN questionnaire
* to evaluate the ability of th FACE PAIN questionnaire to detect change in symptoms following medical or surgical treatment
* to quantify a minimally important difference in the FACE PAIN instrument by correlating disease-specific quality of life change (Transition Scale) with FACE PAIN rating changes following treatment.
* to evaluate the correlation between facial pain symptoms described on the FACE PAIN questionnaire with CT scan and endoscopic findings.

The measurements used for the study are: demographics (age, gender and race), contact information (to facilitate mailing of future instruments), Sinonasal Outcome Test-20 (SNOT-20 - a well validated, 20-item measure of rhinosinusitis specific QOL), FAcial and CEphalic PAin INventory (instrument under study) and Translational Quality of Life Form (this transition scale provides a subjective quantification of the degree of change in quality of life from sinusitis); CT scans and nasal endoscopy findings.

Control subjects will complete the SNOT-20 (validated QOL form) and the FACE PAIN a single time.

Case subjects will complete the SNOT-20 and the FACE PAIN questionnaire at the visit during which they review their CT results with the MD. Thereafter, they will complete the FACE PAIN questionaire twice more; at weeks 12 and 14 post that visit. They will also complete the Transition Scale at week 12. These forms will be mailed to the subjects and returned by mail.

We hypothesize that facial pain ratings will correlate moderately with SNOT-20 scores and a transition scale. Higher values are not expected because QOL instruments encompass many symptoms of chronic sinusitis, but the FACE PAIN instrument addresses location and severity of pain.

We will also test the hypothesis that facial pain ratings will be much lower in non-sinusitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Case subjects from the Rhinology Clinic must have CT evidence of chronic sinusitis
* Control subject from the Otology Clinic who have not had sinus surgery in the past 2 months

Exclusion Criteria:

* any subject unable to give informed consent of complete self-administered questionnaires written in English
* Control subjects with a history of sinusitis in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Rhinology Clinic with a complaint of facial pain and evidence of chronic sinusitis. Control subjects will be patients presenting to the Otology Clinic with no evidence of sinusitis.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg E Davis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Rhinology Clinic, Seattle, Washington, United States